CLINICAL TRIAL: NCT00749957
Title: A Multiple-Site, Phase 1/2, Safety and Efficacy Trial of a Recombinant Adeno-associated Virus Vector Expressing RPE65 (rAAV2-CB-hRPE65) in Patients With Leber Congenital Amaurosis Type 2
Brief Title: Phase 1/2 Safety and Efficacy Study of AAV-RPE65 Vector to Treat Leber Congenital Amaurosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beacon Therapeutics (Industry)
Collaborators: Oregon Health and Science University (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGTC-RPE65-002; R01FD003694 (FDA)
Record Dates: First submitted 2008-09-08; First posted 2008-09-10 (Estimated); Results first posted 2016-04-08 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-10

CONDITIONS: Leber Congenital Amaurosis
Keywords: AAV; adeno-associated virus; RPE65; Leber congenital amaurosis; LCA; gene therapy; human gene transfer
MeSH Terms: conditions — Leber Congenital Amaurosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Subjects at least 6 y/o treated with a lower dose of the vector by subretinal injection
  Interventions: Biological: rAAV2-CB-hRPE65
- 2 (Experimental): Subjects at least 6 y/o treated with a higher dose of the vector by subretinal injection
  Interventions: Biological: rAAV2-CB-hRPE65

INTERVENTIONS:
Biological: rAAV2-CB-hRPE65 — Recombinant adeno-associated virus vector expressing RPE65

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of an adeno-associated virus vector expressing RPE65 in patients with Leber congenital amaurosis caused by mutations in the RPE65 gene.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
This will be a non-randomized, open label study. A total of 12 participants will be enrolled into two groups of 6 each. Each participant will receive rAAV2 CB hRPE65 by subretinal injection in one eye on a single occasion. Participants in Group 1 will receive 450 µL at a dosage level of 4 x 10^11 vg/mL containing a total of 1.8 x 10^11 vg of rAAV2-CB-hRPE65. Participants in Group 2 will receive 450 µL at a dosage level of 1.33 x 10^12 vg/mL containing a total of 6 x 10^11 vg of rAAV2-CB-hRPE65. A retinal surgeon will administer the vector by subretinal injection.

Enrollment will begin with Group 1 and will proceed to Group 2 after review of safety data by a Data and Safety Monitoring Committee.

Safety will be monitored by evaluation of ocular and non ocular adverse events and hematology and clinical chemistry parameters. Efficacy will be measured by evaluation of visual fields, visual acuity and electroretinography.

ELIGIBILITY:
Inclusion Criteria:

* Retinal disease consistent with a diagnosis of Leber congenital amaurosis and documented mutations in the RPE65 gene (including null mutations and mutations that code for abnormal RPE65 protein);
* At least 6 years of age;
* Good general health without significant physical examination findings or clinically significant abnormal laboratory results;
* Able to perform tests of visual and retinal function;
* Visual acuity not better than 20/60 and not worse than hand motion in both the treated eye and the fellow eye;
* Visible photoreceptor (outer nuclear) layer on a standard optical coherence tomography (OCT) scan;
* Acceptable hematology, clinical chemistry and urine laboratory parameters;
* For females of childbearing potential, a negative pregnancy test at screening and at baseline, and agreement to use effective contraception for 12 months after administration of rAAV2-CB-hRPE65, for sexual activity that could lead to pregnancy;
* For males of reproductive potential, agreement to use effective contraception for 12 months after administration of rAAV2-CB-hRPE65, for sexual activity that could lead to pregnancy

Exclusion Criteria:

* Pre-existing eye conditions that would preclude the planned surgery or interfere with interpretation of study endpoints or complications of surgery (e.g. glaucoma, corneal or lenticular opacities, or history or retinal detachment);
* Presence of epiretinal membrane on OCT;
* History of immunodeficiency or other medical conditions that might increase the risk of rAAV2-CB-hRPE65 administration;
* Use of anticoagulants or anti-platelet agents within 7 days prior to study agent administration;
* History of allergy or sensitivity to medications planned for use in the peri-operative period;
* For females of childbearing potential, a positive pregnancy test at screening or baseline (within 2 days before rAAV2-CB-hRPE65 administration);
* Females who are breast feeding;
* Use of any investigational agent, or systemic corticosteroids or other immunosuppressive drug(s), within 3 months prior to enrollment;
* Prior receipt of any AAV gene therapy product;
* Any condition which leads the investigator to believe that the participant cannot comply with the protocol requirements or that may place the participant at an unacceptable risk for participation.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06-17 (Actual); Primary Completion 2014-09-23 (Actual); Study Completion 2017-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Timothy Stout, MD, PhD, MBA, Principal Investigator — Casey Eye Institute, Oregon Health & Science University
Locations (2):
- United States (2):
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Casey Eye Institue, Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Background] Acland GM, Aguirre GD, Bennett J, Aleman TS, Cideciyan AV, Bennicelli J, Dejneka NS, Pearce-Kelling SE, Maguire AM, Palczewski K, Hauswirth WW, Jacobson SG. Long-term restoration of rod and cone vision by single dose rAAV-mediated gene transfer to the retina in a canine model of childhood blindness. Mol Ther. 2005 Dec;12(6):1072-82. doi: 10.1016/j.ymthe.2005.08.008. Epub 2005 Oct 14. PMID 16226919
- [Background] Jacobson SG, Boye SL, Aleman TS, Conlon TJ, Zeiss CJ, Roman AJ, Cideciyan AV, Schwartz SB, Komaromy AM, Doobrajh M, Cheung AY, Sumaroka A, Pearce-Kelling SE, Aguirre GD, Kaushal S, Maguire AM, Flotte TR, Hauswirth WW. Safety in nonhuman primates of ocular AAV2-RPE65, a candidate treatment for blindness in Leber congenital amaurosis. Hum Gene Ther. 2006 Aug;17(8):845-58. doi: 10.1089/hum.2006.17.845. PMID 16942444
- [Background] Weleber RG, Pennesi ME, Wilson DJ, Kaushal S, Erker LR, Jensen L, McBride MT, Flotte TR, Humphries M, Calcedo R, Hauswirth WW, Chulay JD, Stout JT. Results at 2 Years after Gene Therapy for RPE65-Deficient Leber Congenital Amaurosis and Severe Early-Childhood-Onset Retinal Dystrophy. Ophthalmology. 2016 Jul;123(7):1606-20. doi: 10.1016/j.ophtha.2016.03.003. Epub 2016 Apr 19. PMID 27102010
- [Derived] Ku CA, Igelman AD, Huang SJ, Bailey ST, Lauer AK, Duncan JL, Weleber RG, Yang P, Pennesi ME. Perimacular Atrophy Following Voretigene Neparvovec-Rzyl Treatment in the Setting of Previous Contralateral Eye Treatment With a Different Viral Vector. Transl Vis Sci Technol. 2024 Jun 3;13(6):11. doi: 10.1167/tvst.13.6.11. PMID 38888288
- [Derived] Pennesi ME, Weleber RG, Yang P, Whitebirch C, Thean B, Flotte TR, Humphries M, Chegarnov E, Beasley KN, Stout JT, Chulay JD. Results at 5 Years After Gene Therapy for RPE65-Deficient Retinal Dystrophy. Hum Gene Ther. 2018 Dec;29(12):1428-1437. doi: 10.1089/hum.2018.014. Epub 2018 Jul 24. PMID 29869534
- See also: Applied Genetic Technologies Corporation home page — http://agtc.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve subjects with DNA sequence-confirmed mutations in RPE65 were enrolled, 10 at the Casey Eye Institute and 2 at the University of Massachusetts, between June 2009 and September 2012.
Groups:
- Lower Dose of rAAV2-CB-hRPE65: Subjects at least 6 y/o administered a lower dose of the rAAV2-CB-hRPE65 vector by subretinal injection
- Higher Dose of rAAV2-CB-hRPE65: Subjects at least 6 y/o administered a higher dose of the rAAV2-CB-hRPE65 vector by subretinal injection
Period: Overall Study
Arm/Group | Lower Dose of rAAV2-CB-hRPE65 | Higher Dose of rAAV2-CB-hRPE65
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lower Dose of rAAV2-CB-hRPE65: Subjects at least 6 y/o treated with a lower dose of the rAAV2-CB-hRPE65 vector by subretinal injection
- Higher Dose of rAAV2-CB-hRPE65: Subjects at least 6 y/o treated with a higher dose of the rAAV2-CB-hRPE65 vector by subretinal injection
- Total: Total of all reporting groups
Arm/Group | Lower Dose of rAAV2-CB-hRPE65 | Higher Dose of rAAV2-CB-hRPE65 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 22 [6 to 39] | 31 [6 to 37] | 31 [6 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Ocular or Non-ocular Adverse Events
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Lower Dose of rAAV2-CB-hRPE65 | Higher Dose of rAAV2-CB-hRPE65
Number analyzed (Participants) | 6 | 6
participants | 6 | 6

2. Secondary Outcome: Participants With Changes in Visual Fields
Description: Improvement in the central 30 degree visual field, measured by static perimetry, at one or more time points after treatment, that was greater than the limit of agreement for baseline values .
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Lower Dose of rAAV2-CB-hRPE65 | Higher Dose of rAAV2-CB-hRPE65
Number analyzed (Participants) | 6 | 6
participants | 3 | 3

3. Secondary Outcome: Participants With Changes in Best Corrected Visual Acuity
Description: Increase in BCVA of 7 or more letters at Year 2 visit compared to average baseline value
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Lower Dose of rAAV2-CB-hRPE65 | Higher Dose of rAAV2-CB-hRPE65
Number analyzed (Participants) | 6 | 6
participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Lower Dose of rAAV2-CB-hRPE65 | Higher Dose of rAAV2-CB-hRPE65
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Dose of rAAV2-CB-hRPE65 (N=6) | Higher Dose of rAAV2-CB-hRPE65 (N=6)
subconjunctival hemorrhage (Eye disorders) | 3 (3) | 5 (5)
ocular hyperemia (Eye disorders) | 3 (3) | 1 (1)
eye inflammation (Eye disorders) | 0 | 3
eye irritation (Eye disorders) | 1 (1) | 1 (1)
eye pain (Eye disorders) | 1 (2) | 0
eye pruritus (Eye disorders) | 0 | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No